CLINICAL TRIAL: NCT03286062
Title: VM110 in Detection of Microscopic Tumors: A Phase I Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GYN-105
Record Dates: First submitted 2017-09-13; First posted 2017-09-18 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer; Pancreatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Multi dose Phase I study with injection of VM110 at 5 dose levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- VM110 (Experimental): Escalating dose of agent VM110 given to patients to visualize occult cancer with laproscopic infra red detect
  Interventions: Combination Product: Agent VM110 and laproscopic infra-red probe

INTERVENTIONS:
Combination Product: Agent VM110 and laproscopic infra-red probe — Patients with evidence of persistent or recurrent ovarian/ pancreatic cancer would be injected with escalating dose of VM110 24 hr prior to laproscopic surgery to collect biopsy sample in white light and by visualizing the cancerous mass using the laproscopic infra red probe

SUMMARY:
A laproscopic imaging tecgnology that uses a synthetic agent to detect ovarian and pancreatic cancers at an early stage so that patients can get treatment early and prevent the disease from advancing to late stage leading to fatality or recurrence.

DETAILED DESCRIPTION:
Current methods of imaging techniques, CT, MRI and PET, fail to detect moderate volume of diffuse intraperitoneal tumor and provide limited functional information. White light laproscopy is capable of detecting small volume disease in only half of patients in clinical remission, missing occult disease in 30% of this patient population. In this study, a synthetic agent VM110 is to be tested for its ability to detect occult ovarian and pancreatic cancers. The agent is cleaved by proteases, cathepsin B, L, and S and plasmin in cancer cells and the fluorescent cleavage product is detected by near infra red imaging probe. High sensitivity of visualizaion of cancer cells can help detect sub-clinical disease otherwise unidentifiable by usual methods.

Primary Objectives

1. To investigate the safety and toxicity of escalating doses of VM110 administered IV prior to laparoscopic surgery.
2. To define the appropriate dose of VM110 for use in future trials.
3. To define the preliminary efficacy: the optimal dose of VM110 in detection of microscopic peritoneal tumor at laparoscopy not visible with standard white light laparoscopy. Areas visible with both standard white light and NIRF light, and areas visible only with NIRF light will be biopsied. Data from pathologic evaluation of these specimens will be used to determine the efficacy of VM110 with respect to its ability to detect occult disease not visible with standard white light

Secondary Objectives

1. Estimate sensitivity and specificity of VM110 detection
2. Perform correlative pharmacologic and histopathological analyses

ELIGIBILITY:
Inclusion Criteria:

1. Patients with known or suspected pancreatic or ovarian carcinoma who will be undergoing clinically appropriate laparoscopic evaluation or treatment. Patients will not undergo laparoscopy solely for the purpose of participation in this trial.
2. Patients must have evidence of disease either through elevation of tumor markers or radiologic evidence of disease
3. Patient may be male or female and of any race / ethnicity.
4. Participation in this trial will not significantly alter pre-surgical, surgical or post-surgical care
5. ECOG PS of 0-1
6. Patients should be free of active infection requiring antibiotics
7. Any therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
8. Patients must have adequate:

   * Renal function: serum creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
   * Hepatic function: Total bilirubin less than or equal to 1.5 x ULN , SGOT and alkaline phosphatase less than or equal to 2.5 x ULN
   * PTT (partial thromboplastin time) ≤ 1x ULN and INR ≤ 1.5 x ULN.
9. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after. Highly effective contraception methods include combination of any two of the following:

   1. Use of oral, injected or implanted hormonal methods of contraception, or;
   2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
   3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
   4. Total abstinence or;
   5. Male/female sterilization
10. Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to randomization. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child-bearing potential.

    a. Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment
11. Age ≥ 18
12. Capable of complying with study procedures and communicating with study personnel.
13. Patients must have signed an approved informed consent and authorization permitting release of personal health information. Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria:

1. Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded. Prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease.
2. Patients with an active bleeding diathesis or on oral anti-vitamin K medication (except low-dose warfarin used for catheter-related thrombosis prophylaxis).
3. Prior history of hypersensitivity to Pegylated liposomal doxorubicin or ICG allergy. Caution should be taken if prior ICG allergy is noted.
4. Pregnant or nursing (lactating) women
5. History of congestive cardiac failure or an EKG suggesting significant conduction defect, or myocardial ischemia, or active psychiatric disease requiring treatment that would interfere with the understanding or conduct of the study.
6. Subject has previously received VM110, or any other investigational product in the past thirty days.
7. Inadequate tumor sites or volume to allow for biopsy per standard of care.
8. Patients with psychiatric or other conditions rendering them incapable of participating in informed consent or the requirements of this protocol or other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete good quality data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of VM110 related toxicity assessed by NCI CTCAE criteria 4.03 | 3-62 weeks
  Patients would be monitored for severity of adverse events due to VM110 based on NCI CTCAE criteria 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Gina Martina-Smaldone, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No